CLINICAL TRIAL: NCT06355102
Title: The Generation and Chronicity of Tinnitus in Patients With Sudden Sensorineural Hearing Loss: Insights From fMRI and Serum Metabolomics Analysis
Brief Title: The Development of Tinnitus in Patients With SSNHL: Insights From fMRI and Metabolomics
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-116
Record Dates: First submitted 2024-03-12; First posted 2024-04-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sudden Sensorineural Hearing Loss; Tinnitus
Keywords: Sudden sensorineural hearing loss; Tinnitus chronicity; Functional magnetic resonance imaging; Metabolomics
MeSH Terms: conditions — Hearing Loss, Sudden; Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study collects serum samples from subjects for the purpose of serum metabolomics research, and relevant samples will be destroyed after the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SSNHL with Tinnitus: Patients diagnosed with sudden sensorineural hearing loss accompanied with acute occuring tinnitus symptoms.
  Interventions: Other: Conventional treatment and care
- SSNHL without Tinnitus: Patients diagnosed with sudden sensorineural hearing loss without acute occuring tinnitus symptoms.
  Interventions: Other: Conventional treatment and care
- Health Control: Healthy subjects with normal hearing and no tinnitus.
  Interventions: Other: Conventional treatment and care

INTERVENTIONS:
Other: Conventional treatment and care — Conventional treatment and care

SUMMARY:
The goal of this clinical trial is to investigate the factors and mechanisms underlying tinnitus generation and chronification in patients with sudden sensorineural hearing loss (SSNHL) . The main questions it aims to answer are:

* What are the peripheral and central influencing factors that contribute to tinnitus in patients with SSNHL?
* Can serum metabolic biomarkers be identified to predict and monitor tinnitus prognosis in these patients?

Participants in this study will include patients with SSNHL and tinnitus, patients with SSNHL without tinnitus, and healthy subjects. They will be asked to undergo a series of assessments, including audiological tests, vestibular function examinations, and functional magnetic resonance imaging (fMRI). Additionally, blood samples will be collected for metabolomics analysis.

Investigators will compare the brain functional states and serum metabolite profiles of patients with SSNHL and tinnitus to those without tinnitus. Morever, tinnitus symptom characteristics, audiological outcomes, and brain functional states will be assessed during time.

DETAILED DESCRIPTION:
The incidence rate of tinnitus is very high globally and shows an increasing trend year by year. Sudden sensorineural hearing loss (SSNHL) , a prevalent otolaryngological emergency, often coincides with tinnitus among its patient population. This condition can significantly impact individuals' interpersonal relationships, work performance, and daily functioning, ultimately leading to a diminished quality of life and even psychological disturbances, such as anxiety and depression. Consequently, it is imperative to expore the mechanisms underlying the emergence and chronicity of tinnitus following SSNHL, and to devise targeted intervention strategies aimed at preventing the chronicity of tinnitus.

This study aims to enroll 30 patients with SSNHL accompanied by tinnitus, 30 patients with SSNHL without tinnitus, and 30 healthy subjects. Investigators will record general demographic information, tinnitus symptom characteristics, audiological examinations, vestibular function tests, and other information for each group during the acute phase of SSNHL onset. Using functional magnetic resonance imaging (fMRI), investigators will compare the brain functional states of patients with SSNHL accompanied by tinnitus and those without tinnitus during the acute phase to investigate the peripheral influencing factors and central mechanisms of tinnitus production. Additionally, investigators will conduct metabolomics analysis to compare the serum metabolite profiles of these two patient groups to identify serum metabolic biomarkers and prognostic biomarkers for tinnitus in patients with SSNHL accompanied by tinnitus. Furthermore, this study will conduct follow-up assessments on the subjects at 1 month, 3 months, and 6 months after the onset of SSNHL, reviewing changes in their symptom characteristics, audiological examinations, and fMRI. At 6 months after the onset, patients will be divided into a tinnitus recovery group and a tinnitus non-recovery group based on their tinnitus recovery status. Investigators will compare the general demographic characteristics, audiological examinations, and brain functional MRI findings between the two groups to explore the role and mechanisms of brain plasticity changes in the recovery or chronicity of tinnitus in patients with SSNHL.

ELIGIBILITY:
Inclusion Criteria:

1. Group of SSNHL with Tinnitus:

   1. Age between 18 and 65 years old;
   2. Meets the diagnostic criteria for SSNHL; untreated within 5 days after onset;
   3. Presence of tinnitus;
   4. Able to complete questionnaires independently and cooperate with fMRI and follow-up assessments.
2. Group of SSNHL without Tinnitus:

   1. Age between 18 and 65 years old;
   2. Meets the diagnostic criteria for SSNHL; untreated within 5 days after onset;
   3. Absence of tinnitus;
   4. Able to complete questionnaires independently and cooperate with fMRI and follow-up assessments.
3. Healthy Control:

   1. Age between 18 and 65 years old;
   2. Normal hearing screening results;
   3. Able to complete questionnaires independently and cooperate with fMRI and follow-up assessments.

Exclusion Criteria:

1. Previous diagnosis of otic organic diseases such as otitis media, cholesteatoma of the middle ear, Ménière's disease, acoustic neuroma, hereditary deafness, inner ear malformations, etc.; history of ear surgery; long-term exposure to noise; use of ototoxic drugs;
2. Presence of brain organic diseases such as cerebral infarction, brain tumor, or contraindications for functional magnetic resonance imaging (fMRI) during nuclear magnetic resonance (NMR) examination;
3. History of mental illness, including anxiety, depression, insomnia, etc.;
4. Individuals unable to cooperate due to severe mental factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SSNHL and individuals undergoing physical examination at the Department of Otolaryngology, the First Affiliated Hospital of Nanjing Medical University
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Brain function states | Acute phase (within 5 days after onset), 1 month, 3 months, and 6 months after onset
  Fractional amplitude of low-frequency fluctuation, regional homogeneity, and functional connection will be compared among different groups using fMRI. Morever, the connections between the default mode network (DMN), central executive network (CEN), and salience network (SN) will be assessed through fMRI.
Serum metabolomics | Acute phase (within 5 days after onset)
  Serum metabolic profiles and characteristics will be gained and compared in patients SSNHL with or with tinnitus, using LC-MS metabolomics technology.

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhang, M.D., Principal Investigator — Department of Otolaryngology, the First Affiliated Hospital, Nanjing Medical University
Locations (1):
- Department of Otolaryngology, the First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China